CLINICAL TRIAL: NCT00859547
Title: A Phase 4, Open-Label, Single-Group Safety and Immunogenicity Study of RECOTHROM® (rThrombin) in Pediatric Subjects Undergoing Synchronous Burn Wound Excision and Skin Grafting
Brief Title: Safety and Immunogenicity Study of Recombinant Thrombin (rThrombin) in Pediatric Participants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ZymoGenetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 499H01
Record Dates: First submitted 2009-03-09; First posted 2009-03-11 (Estimated); Results first posted 2011-12-08 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Blood Loss, Surgical
MeSH Terms: conditions — Blood Loss, Surgical | interventions — recombinant human thrombin; Thrombin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Recombinant thrombin (rThrombin), 1000 IU/mL (Experimental)
  Interventions: Biological: rThrombin, 1000 IU/mL

INTERVENTIONS:
Biological: rThrombin, 1000 IU/mL — rThrombin,1000 IU/mL, 1000 IU/mL, applied topically to the bleeding site during a single surgery procedure on Day 1.
  Other Names: RECOTHROM

SUMMARY:
The objective of this study is to assess the safety and immunogenicity of recombinant thrombin (rThrombin) administered as an aid to hemostasis during burn wound excision and skin grafting in pediatric patients, newborn through 17 years of age.

DETAILED DESCRIPTION:
The safety, immunogenicity, and efficacy of rThrombin have been evaluated in 5 Phase 2 studies, 1 pivotal Phase 3 study, and 1 Phase 3b study, in surgical indications such as: spinal surgery, major hepatic resection, peripheral arterial bypass surgery, arteriovenous graft formation for hemodialysis access, and burn wound excision. Limited data currently exist on the effects of rThrombin exposure in pediatric patients. This Phase 4 trial aims to provide additional information on the use of rThrombin in children by evaluating the drug's safety and immunogenicity when administered as an aid to hemostasis during burn wound excision and skin grafting in pediatric burn patients.

ELIGIBILITY:
Inclusion Criteria:

* Age of newborn through 17 years at time of enrollment
* At least 1 skin graft recipient site measuring at least 1% of total body surface area (TBSA)
* Total initial burn wounds estimated to measure less than 40% of TBSA
* Bleeding indicating treatment with rThrombin during the surgical procedure
* Females of child-bearing potential must have a negative urine or serum pregnancy test within 2 days prior to study-drug treatment
* informed consent document signed by legal representative (guardian) and approved by an institutional review board/independent ethics committee (IRB/IEC)
* Participant has signed an IRB/IEC-approved pediatric assent document, if applicable

Exclusion Criteria:

* Gestational age younger than 36 weeks at birth (for infants younger than 2 years)
* Documented active infection at the graft recipient site (participants with resolved infections at potential graft recipient sites are not excluded)
* Acute inhalation injury, as defined by bronchoscopic evidence of lower airway injury
* Currently undergoing autologous skin grafting for ischemic ulcer disease or cutaneous malignancies
* Presence of antibodies or hypersensitivity to the study drug or any of its components, other thrombin preparations, or coagulation factors
* Transfusion of whole blood, fresh frozen plasma, cryoprecipitate, or platelets within 24 hours prior to study-drug treatment (packed red blood cell transfusions are allowed)
* History of HIV infection or other immunodeficiency syndrome or is taking immunosuppressive or antirejection medications
* Medical, social, or psychosocial factors that, in the opinion of the investigator, could affect safety or compliance with study procedures
* Breastfeeding or being breastfed
* Treatment with any experimental agent within 30 days of study enrollment or treatment

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2009-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Foster, MD, Principal Investigator — Arizona Burn Center
Locations (1):
- Arizona Burn Center, Phoenix, Arizona, United States

REFERENCES:
- [Derived] Sinha S, Gabriel VA, Arora RK, Shin W, Scott J, Bharadia SK, Verly M, Rahmani WM, Nickerson DA, Fraulin FO, Chatterjee P, Ahuja RB, Biernaskie JA. Interventions for postburn pruritus. Cochrane Database Syst Rev. 2024 Jun 5;6(6):CD013468. doi: 10.1002/14651858.CD013468.pub2. PMID 38837237
- [Derived] Foster KN, Mullins RF, Greenhalgh DG, Gamelli RL, Glat P, Lentz CW, Kahn SA, Brandigi C, Fredlund P, Alexander WA. Recombinant human thrombin: safety and immunogenicity in pediatric burn wound excision. J Pediatr Surg. 2011 Oct;46(10):1992-9. doi: 10.1016/j.jpedsurg.2011.05.022. PMID 22008340

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 32 participants who signed informed consent in this study, 30 were actually enrolled and received treatment with rThrombin.
Groups:
- rThrombin, 1000 IU/mL: Recombinant thrombin (rThrombin), 1000 IU/mL, applied topically during a single surgery procedure on Day 1.
Period: Overall Study
Arm/Group | rThrombin, 1000 IU/mL
Started | 30
Completed | 28
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Parent withdrew consent | 1

BASELINE CHARACTERISTICS:
Arm/Group | rThrombin, 1000 IU/mL
Number analyzed (Participants) | 30
Age, Customized [Number; unit: participants]
  0-2 years | 11
  3-6 years | 8
  7-11 years | 3
  12-17 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian/Alaskan native | 1
  Black or African American | 6
  Hispanic | 9
  White | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Death, Serious Adverse Events, Treatment-related Adverse Events (AE), AEs Leading to Discontinuation, and AEs of Hypersensitivity
Description: An AE is any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not necessarily have a causal relationship with treatment. An SAE is any unfavorable medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency or abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=possibly, probably, or certainly related to and of unknown relationship to study treatment
Time Frame: Days 1 through 29, continuously
Population: Participants who received treatment with rThrombin.
Measure: Number; unit: Participants
Arm/Group | rThrombin, 1000 IU/mL
Number analyzed (Participants) | 30
Participants
  Deaths | 0
  Serious adverse events | 1
  Treatment-related adverse events (AEs) | 0
  AEs leading to discontinuation | 0
  AEs of hypersensitivity | 3

2. Primary Outcome: Number of Participants With AEs by Maximum Severity
Description: An AE is any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not necessarily have a causal relationship with treatment. Mild=asymptomatic or minor symptoms; intervention not indicated. Moderate=requiring only minimal, local, or noninvasive intervention. Severe=significant symptoms but not life-threatening; hospitalization or invasive intervention indicated. Life-threatening=indicating intensive care or urgent invasive intervention.
Time Frame: Days 1 through 29, continuously
Population: Participants who received treatment with rThrombin.
Measure: Number; unit: Participants
Arm/Group | rThrombin, 1000 IU/mL
Number analyzed (Participants) | 30
Participants
  Mild (0-2 years, n=11) | 3
  Mild (3-6 years, n=8) | 3
  Mild (7-11 years, n=3) | 0
  Mild (12-17 years, n=8) | 3
  Moderate (0-2 years, n=11) | 1
  Moderate (3-6 years, n=8) | 5
  Moderate (7-11 years, n=3) | 3
  Moderate (12-17 years, n=8) | 3
  Severe (0-2 years, n=11) | 3
  Severe (3-6 years, n=8) | 0
  Severe (7-11 years, n=3) | 0
  Severe (12-17 years, n=8) | 1
  Life-threatening (0-2 years, n=11) | 3
  Life-threatening (3-6 years, n=8) | 0
  Life-threatening (7-11 years, n=3) | 0
  Life-threatening (12-17 years, n=8) | 0

3. Secondary Outcome: Number of Participants WIth Positive Findings for Anti-rThrombin Product Antibody
Description: Antibody-positive was defined as seroconversion or ≥1.0 unit (≥10-fold) increase in titer compared with antibody titer at baseline.
Time Frame: At Day 29
Population: Participants who received study drug and had both baseline and on-treatment anti-rThrombin product antibody assessments.
Measure: Number; unit: Participants
Arm/Group | rThrombin, 1000 IU/mL
Number analyzed (Participants) | 27
Participants | 0

4. Primary Outcome: Number of Participants With Clinical Laboratory Findings of Grade O or Higher in Platelet, White Blood Cell (WBC), Lymphocyte, and Neutrophil Counts
Description: Abnormal laboratory findings were recorded as AEs when considered clinically significant (unusual for the surgical population or individual participant) by the investigator, when associated with symptoms, when requiring specific treatment, or when requiring a change in participant management.LLN=lower level of normal. Platelets: Grade 0=normal. WBC: Grade 0=normal. Lymphocytes: Grade 0=normal; Grade 1=<LLN x 0.8-10^9/L. Neutrophils: Grade 0=normal; Grade 1=<LLN-1.5x10^9/L; Grade 2=<1.5-1.0x10^9/L
Time Frame: Baseline and Day 29 from Baseline
Population: Participants who received treatment with rThrombin.
Measure: Number; unit: Participants
Arm/Group | rThrombin, 1000 IU/mL
Number analyzed (Participants) | 30
Participants
  Grade 0, low platelets (Baseline) | 30
  Grade 0, low platelets (Day 29, N=25) | 25
  Grade 0, low WBC (Baseline) | 30
  Grade 0, low WBC (Day 29, N=26) | 26
  Grade 0, low lymphocytes (Baseline, N=29) | 28
  Grade 0, low lymphocytes (Day 29, N=25) | 25
  Grade 1, low lymphocytes (Baseline, N=29) | 1
  Grade 1, low lymphocytes (Day 29, N=25) | 0
  Grade 0, neutrophils (Baseline, N=29) | 29
  Grade 0, neutrophils (Day 29, N=25) | 24
  Grade 2, low neutrophils (Baseline) | 0
  Grade 2, low neutrophils (Day 29, N=25) | 1

5. Primary Outcome: Number of Participants With Clinical Laboratory Findings of Grade 0 or Higher in Hemoglobin Levels
Description: LLN=lower level of normal. Grade 1=100 g/L to <LLN; Grade 2=80 to <100 g/L; Grade 3=65 to <80 g/L; Grade 4=<65 g/L.
Time Frame: Baseline and Day 29 from Baseline
Population: Participants who received treatment with rThrombin.
Measure: Number; unit: Participants
Arm/Group | rThrombin, 1000 IU/mL
Number analyzed (Participants) | 30
Participants
  Grade 1 low hemoglobin (Baseline) | 13
  Grade 1 low hemoglobin (Day 29, N=26) | 7
  Grade 2 low hemoglobin (Baseline) | 4
  Grade 2 low hemoglobin (Day 29, N=26) | 5
  Grade 3 low hemoglobin (Baseline) | 1
  Grade 3 low hemoglobin (Day 29, N=26) | 0
  Grade 4 low hemoglobin (Baseline) | 0
  Grade 4 low hemoglobin (Day 29, N=26) | 0

6. Primary Outcome: Number of Participants With Clinical Laboratory Findings of Grade 0 or Higher in Creatinine Levels
Description: ULN=upper level of normal. Grade 0=normal; Grade 1=>ULN to 1.5 x ULN.
Time Frame: Baseline and Day 29 from Baseline
Population: Participants who received treatment with rThrombin.
Measure: Number; unit: Participants
Arm/Group | rThrombin, 1000 IU/mL
Number analyzed (Participants) | 30
Participants
  Grade 0 high creatinine (Baseline, N=30) | 30
  Grade 0 high creatinine (Day 29, N=26) | 25
  Grade 1 high creatinine (Baseline) | 0
  Grade 1 high creatinine (Day 29, N=26) | 1

7. Primary Outcome: Number of Participants With Elevations in the Coagulation Parameter of Activated Partial Thromboplastin Time (aPPT)of Grade 0 or Higher
Description: ULN=upper limit of normal. Grade 0=normal; Grade 1=ULN to 1.5 x ULN.
Time Frame: Baseline and Day 29 from Baseline
Population: Participants who received treatment with rThrombin.
Measure: Number; unit: Participants
Arm/Group | rThrombin, 1000 IU/mL
Number analyzed (Participants) | 29
Participants
  Grade 0 high aPPT (Baseline, N=29) | 22
  Grade 0 high aPPT (Day 29, N=24) | 19
  Grade 1 high aPPT (Baseline, N=29) | 7
  Grade 1 high aPPT (Day 29, N=24) | 5

8. Primary Outcome: Number of Participants With a High International Normalized Ratio (INR) of Prothrombin Time of Grade 0 or Higher
Description: Grade 0=normal.
Time Frame: Baseline and Day 29 from Baseline
Population: Participants who received treatment with rThrombin.
Measure: Number; unit: Participants
Arm/Group | rThrombin, 1000 IU/mL
Number analyzed (Participants) | 28
Participants
  Grade 0 INR High (Baseline, N=28) | 28
  Grade 0 INR High (Day 29, N=24) | 24

ADVERSE EVENTS:
Arm/Group | TOTAL
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 28/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TOTAL (N=30)
TRANSPLANT REJECTION (Immune system disorders) | 1
SKIN GRAFT INFECTION (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TOTAL (N=30)
ANAEMIA (Blood and lymphatic system disorders) | 9
CONSTIPATION (Gastrointestinal disorders) | 2
VOMITING (Gastrointestinal disorders) | 2
OEDEMA PERIPHERAL (General disorders) | 2
PYREXIA (General disorders) | 3
TRANSPLANT REJECTION (Immune system disorders) | 3
BACTERAEMIA (Infections and infestations) | 2
SKIN GRAFT INFECTION (Infections and infestations) | 2
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 15
SEROMA (Injury, poisoning and procedural complications) | 2
SKIN GRAFT FAILURE (Injury, poisoning and procedural complications) | 2
WOUND SECRETION (Injury, poisoning and procedural complications) | 2
EXCESSIVE GRANULATION TISSUE (Skin and subcutaneous tissue disorders) | 2
PRURITUS (Skin and subcutaneous tissue disorders) | 13
HAEMATOMA (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
ZymoGenetics (ZG) agreements vary by trial, but each states that presentation/publication (p/p) cannot disclose Confidential Information (CI), excluding trial results; p/p may not begin until the earlier of 18 months after study end, ZG/lead investigator publishes, or ZG notification that multicenter publication is not planned; ZG has specified time for draft review before submission/presentation and may delay or modify content, require CI removal, and delay p/p for patent application filing.